CLINICAL TRIAL: NCT05024396
Title: Validity and Reliability of Jump Height in Healthy Athletic Persons Measured With a Sensor
Brief Title: Validity and Reliability of Jump Height
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-D0004
Record Dates: First submitted 2021-07-22; First posted 2021-08-27 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- maximum jump height (Experimental): Two visits will take place 1-2 weeks apart. At the first visit, participants will complete 2x3 single-leg countermovement jumps measured by two subjects each. At the second visit, three jumps are completed measured by the first test subject.
  Interventions: Diagnostic Test: maximum jump height

INTERVENTIONS:
Diagnostic Test: maximum jump height — Three single leg countermovement jumps were performed. The maximum jump height is measured with a sensor that is adapted at the subjects'leg and with a force plate.

SUMMARY:
The primary objective is to test intratester and intertester reliability of maximum jump height using the sensor Orthelligent Pro.

The secondary objective is to test the concurrent validity of maximum jump height measured with the Orthelligent Pro compared to the gold standard which is the force plate.

DETAILED DESCRIPTION:
In everyday physiotherapy practice, there is often no budget for expensive measuring instruments. Thus, devices such as a force plate are rarely available. Physiotherapists are always looking for inexpensive, practical and portable measuring instruments to evaluate therapy outcomes and to make reliable statements about the time for Return to Sport. Maximum jump height is a performance-determining factor in various jump-intensive game sports. In addition, the jump height serves as an important criterion to decide when an athlete can return to his usual sport after an injury. There is a new sensor on the market that measures jump height. This sensor is called Orthelligent Pro. It is shown to be a cost-effective and feasible measurement method for return to sport in physical therapy practice. So far, validity and reliability has never been tested. Therefore, this study aims to test the validity and reliability of the Orthelligent Pro for the measurement of maximum jump height. Two visits will take place 1-2 weeks apart. At the first visit, participants will complete 2x3 single-leg countermovement jumps measured by two testers each. At the second visit, three jumps are completed measured by the first tester.

The primary objective is to evaluate the intra-and intertester reliability of maximum jump height using Orthelligent Pro. The secondary objective is to test the concurrent validity of maximum jump height measured with the Orthelligent Pro compared with the gold standard which is the force plate. The primary and secondary endpoints are maximum jump height measured in centimeters.

ELIGIBILITY:
Inclusion Criteria:

* male and female persons aged 18-65 years
* performing at least 1x / week a training including jumping elements
* familiar with counter movement jumps
* good knowledge of German
* understand verbal and written instructions
* signed informed consent

Exclusion Criteria:

* known pregnancy
* known or suspected non-compliance with the protocol
* drug or alcohol abuse
* inability of the individual to follow the testing procedures, e.g., due to language problems, mental illness, dementia, etc.
* injuries of the lower extremity in the past year
* concomitant diseases of the foot, knee or hip
* tiring activity of the lower extremity the day before the test
* vigorous activity of the lower extremity one hour before the test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
maximum jump height | two weeks
  the maximum jump height will be measured in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Pasquale, Principal Investigator — University of Zurich
Locations (1):
- Physiotherapie Occupational Therapy University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No